CLINICAL TRIAL: NCT05242874
Title: Anti-emetic Prophylaxis Using Fosaprepitant , Tropisetron, and Olanzapine, With or Without Dexamethasone for Anthracycline and Cyclophosphamide Chematherapy: A Multicenter, Randomized, Open-labeled Phase 3 Trial
Brief Title: Anti-emetic Prophylaxis With or Without Dexamethasone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Director, Head of Breast Oncology, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HELEN-009
Record Dates: First submitted 2022-01-28; First posted 2022-02-16 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: Nausea; Vomiting; Glucocorticoids; Olanzapine; Tropisetron; Fosaprepitant; Signs and Symptoms, Digestive; Antiemetics; Physiological Effects of Drugs
MeSH Terms: conditions — Vomiting; Nausea; Signs and Symptoms, Digestive | interventions — fosaprepitant; Tropisetron; Olanzapine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triple group (Experimental): A three-drug antiemetic regimen with fosaprepitant, tropisetron, and olanzapine (triple group)
  Interventions: Drug: Fosaprepitant, tropisetron, and olanzapine-based antiemetic regimen
- Quadruple group (Active Comparator): A four-drug regimen including fosaprepitant, tropisetron, olanzapine, and dexamethasone (quadruple group)
  Interventions: Drug: Fosaprepitant, tropisetron, olanzapine, and dexamethasone-based antiemetic regimen

INTERVENTIONS:
Drug: Fosaprepitant, tropisetron, and olanzapine-based antiemetic regimen — Fosaprepitant 150 mg intravenously on Day 1, tropisetron 5 mg intravenously on Day 1, and olanzapine 5 mg orally on Days 1 to 4.
  Other Names: Fosaprepitant+Tropisetron+Olanzapine
  Arms: Triple group
Drug: Fosaprepitant, tropisetron, olanzapine, and dexamethasone-based antiemetic regimen — Fosaprepitant 150 mg intravenously on Day 1, tropisetron 5 mg intravenously on Day 1, and olanzapine 5 mg orally on Days 1 to 4. Dexamethasone 12 mg on Day 1, followed by 8 mg on Days 2 to 4.
  Other Names: Fosaprepitant+Tropisetron+Olanzapine+Dexamethasone
  Arms: Quadruple group

SUMMARY:
To evaluate the efficacy and safety of a fosaprepitant, tropisetron, and olanzapine antiemetic regimen, with or without dexamethasone, in patients receiving highly emetogenic chemotherapy with epirubicin and cyclophosphamide.

DETAILED DESCRIPTION:
Patients in this study were randomly assigned in a 1:1 ratio to one of two groups using an interactive response system with permuted blocks of four, stratified by age (<55 vs. ≥55 years). They received either a three-drug antiemetic regimen with fosaprepitant, tropisetron, and olanzapine (triple group) or a four-drug regimen including fosaprepitant, tropisetron, olanzapine, and dexamethasone (quadruple group). All patients were hospitalized for approximately 120 hours post-chemotherapy, documenting emetic episodes, rescue medication use, and nausea ratings on a Likert scale (0 = no nausea, 1 = mild nausea, 2 = moderate nausea, 3 = severe nausea) in a diary. Rescue therapy was available as needed. Clinical staff monitored adverse events every 24 hours using National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. Subjects who initiated treatment were followed up for endpoints, including complete response (CR), complete control (CC), total control (TC), quality of life, and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer patients receiving their first anthracycline/cyclophosphamide-based HEC regimen (cyclophosphamide 600 mg/m², epirubicin 90-100 mg/m²); divided doses excluded.
2. No prior chemotherapy.
3. Aged 18-70 years.
4. ECOG performance status 0 or 1.
5. Adequate organ function: (including absolute neutrophil count≥1,500/mm3, WBC count≥3,000/mm3, platelet count≥100,000/mm3, AST< 2.5×the upper limit of normal (ULN), ALT< 2.5×ULN, bilirubin< 1.5×ULN, creatinine< 1.5×ULN).
6. No nausea or vomiting within 24 hours before registration.
7. Negative pregnancy test within 7 days prior (women of childbearing potential).
8. No severe cognitive impairment.
9. No hypersensitivity to fosaprepitant, tropisetron, olanzapine, and dexamethasone.
10. No significant cardiac issues: arrhythmia, recent heart failure, or myocardial infarction within 6 months.
11. No symptomatic brain metastasis or carcinomatous meningitis.
12. No diabetes requiring insulin or oral medication.
13. No use of prohibited medications within 48 hours before registration or during treatment.
14. Informed consent obtained.

Exclusion Criteria:

1. History of allergic reactions to study drugs or their analogues.
2. Nausea and vomiting requiring antiemetic treatment at registration.
3. Pregnant or nursing women, those who may become pregnant, or those not planning to use contraception.
4. Mental illness or psychiatric symptoms interfering with daily activities, making study participation difficult.
5. Diabetes treated with insulin/oral hypoglycemics or HbA1c (NGSP) ≥ 6.5% or HbA1c (JDS) ≥ 6.1% at registration.
6. Recent (within 6 months) unstable angina, myocardial infarction, cerebral hemorrhage, cerebral infarction, or active gastroduodenal ulcer.
7. Convulsive disorders requiring anticonvulsants, ascites needing therapeutic puncture, or gastrointestinal obstruction.
8. Inability to be hospitalized for up to 120 hours (Day 6) post-AC administration initiation.
9. Any other conditions deemed inappropriate for study participation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Complete response rate (CR) during overall (0-120 hours after the initiation of anthracycline/cyclophosphamide administration) phase. | 0-120 hours after the initiation of anthracycline/cyclophosphamide administration
  CR was determined by the absence of any retching or vomiting and the absence of any requirement for additional antiemetic treatment.

SECONDARY OUTCOMES:
CR during the acute (0-24 hours after the initiation of anthracycline/cyclophosphamide administration) and delayed (24-120 hours after the initiation of anthracycline/cyclophosphamide administration) phase | 0-24 hours and 24-120 hours after the initiation of anthracycline/cyclophosphamide administration
  CR was determined by the absence of any retching or vomiting and the absence of any requirement for additional antiemetic treatment.
Complete control rate (CC) during the acute, delayed, and overall phase | Day 1 to day 5 after the initiation of anthracycline/cyclophosphamide administration
  CC is defined as a condition in which a patient does not report more than mild nausea (0 or 1 on a 4-grade categorical scale) (0 = no nausea, 1 = mild nausea, 2 = moderate nausea, 3 = severe nausea).
Total control rate (TC) during the acute, delayed, and overall phases | Day 1 to day 5 after the initiation of anthracycline/cyclophosphamide administration
  TC is defined as a condition in which a patient does not report any nausea (0 on a 4-grade categorical scale) (0 = no nausea, 1 = mild nausea, 2 = moderate nausea, 3 = severe nausea).
Safety outcomes | Day 1 to day 5 after the initiation of anthracycline/cyclophosphamide administration
  Adverse event incidence rate
Quality of life based on Functional Living Index-Emesis (FLIE) assessment | 0-120 hours after the initiation of anthracycline/cyclophosphamide administration
  Quality of life based on Functional Living Index-Emesis (FLIE) assessment in the overall phase (0-120 h).
Exploratory endpoints-The time to the treatment failure | 0-120 hours after the initiation of anthracycline/cyclophosphamide administration
  The time to the treatment failure (time to ﬁrst emetic episode or time to ﬁrst use of rescue medication, whichever occurred ﬁrst).

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhen Liu, Principal Investigator — Henan Cancer Hospital
Locations (2):
- China (2):
  - Henan cacer hospital, Henan, Henan
  - Henan cancer hospital, Zhengzhou, Henan